CLINICAL TRIAL: NCT00211848
Title: Antiviral & Antifibrotic Liver Therapy in HCV + Drinkers and Non-Drinkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AA12867; 99-1097
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2007-04

CONDITIONS: Hepatitis C
Keywords: Chemical Compounds-drugs; Human Subjects- adults; Gastrointestinal System-liver; Pathology
MeSH Terms: conditions — Hepatitis C | interventions — lipostabil; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Polyenylphosphatidylcholine (PPC)
Drug: Pegylated Interferon
Drug: Ribavirin

SUMMARY:
The primary aim of this investigation is to evaluate the effect of a combined antiviral, antifibrotic and antioxidant treatment on the progression of liver disease in patients with hepatitis C who either abstain from alcohol or continue to drink. All subjects are given state-of-the-art antiviral treatment (pegylated interferon + ribavirin), supplemented with either placebo or polyenylphosphatidylcholine (PPC), a purified soybean extract consisting of 95-96% polyunsaturated phosphatidylcholines (PC) and which has both antifibrotic and antioxidant properties. Secondary aims are to verify whether moderate alcohol consumption interferes with the antiviral effect of pegylated interferon + ribavirin on HCV and to validate the reliability of various circulating markers as substitute for liver biopsies to indicate the stage of liver pathology and its propensity for progression.

DETAILED DESCRIPTION:
Current therapy for HCV disease focuses on anti-viral treatment. The combination of pegylated interferon and ribavirin is approved by the FDA for treating HCV disease. Subjects in this study will be given ribavirin and pegylated interferon. One innovative aspect of this proposal is that the state-of-the-art antiviral treatment will be supplemented by an anti-fibrotic agent, namely polyenylphosphatidylcholine (PPC), or placebo, administered in a double blind randomized fashion. Current therapy focuses on anti-viral treatment, neglecting the fact that what causes the medical symptoms and eventually the demise of the HCV patient is the liver fibrosis, the resulting cirrhosis and the associated complications, including hepatocellular carcinoma. If the fibrotic process could be stopped or even prevented, the hepatitis C virus would lose much of its impact on health. Available anti-fibrotic agents are too toxic to be used in patients, except for one, namely PPC, which has been shown in various experimental models to have striking anti-fibrotic actions, and was found recently, in a European study, to be beneficial in patients with hepatitis C in terms of their circulating levels of transaminases. Various studies have indicated that HCV is associated with an oxidative stress and thus it is noteworthy that PPC was discovered to have also significant anti-oxidant effects.

The study has been approved by the Institutional Review Board at each Center, and all the patients are provided written informed consent. After screening, patients are randomly assigned to one of 2 treatment groups (PPC or placebo). The two treatment groups are given the combination of pegylated interferon (180 μg injected once weekly) (Shiffman et al, 1999; Sulkowski et al, 1999), and ribavirin for 48 weeks (genotype I) or 24 weeks (other genotypes). If the latter do not respond in terms of HCV RNA, they are also treated for 48 weeks. Ribavirin is administered orally twice a day at a total daily dose of 1000 mg for patients who weigh 75 kg or less and 1200 mg for those who weigh more than 75 kg. These drugs are started and stopped at the same time, the PPC (5 chewable tablets of 0.9 gm each per day) or corresponding placebo (obtained from PHOSPHOLIPID GmbH, a successor of Rhone-Poulenc Rorer, Cologne, Germany) are given to each patient for the 3 years.

The patients in whom the hemoglobin falls by more than 2 g per deciliter are followed every 2 weeks until stabilization. The dose of ribavirin is reduced to 600 mg per day in patients whose hemoglobin concentrations fall below 10 g per deciliter, and it is discontinued if the concentration falls below 8.5 g per deciliter. For severe adverse events other than anemia, the dose of interferon is reduced in half and the dose of ribavirin to 600 mg per day. The full dose can be resumed after the event, or discontinued if the effect persists.

The patients are evaluated as outpatients at weeks 1, 2, 4 and then every 4 weeks during the 24-48 weeks of interferon-ribavirin-PPC (or placebo) treatment as well as during the subsequent PPC (placebo) therapy. Upon cessation of antiviral treatment, study patients may be seen on a quarterly basis if, in the Investigator's judgment, this flexible schedule will not impact negatively on patient care but will impact positively on patient retention. Biochemical testing is performed by a central laboratory. Plasma HCV RNA levels are determined before treatment, during interferon-ribavirin treatment at 24 and 48 weeks, after interferon-ribavirin therapy at months 18, 24 and 30 and at the end of the 3 years. Plasma HCV RNA is measured by a quantitative reverse-transcription-polymerase-chain-reaction assay (Cobas Amplicor for HCV Monitor v.2, Roche Diagnostic Systems, Inc.) that has a sensitivity of 3000 IU/ml with a linearity up to 2.5 X 106 IU/ml. Samples negative with the quantitative HCV-RNA are retested with the qualitative HCV-PCR assay (Cobas Amplicor for HCV 2.0, Roche Diagnostic Systems, Inc.) that has a sensitivity of 60 IU/ml. HCV genotyping is carried out according to Stuyver et al, (1993; Inno-LIPA HCVII, Immunogenetics).

Compliance in terms of PPC (or placebo) will be monitored by 4 methods: patient diary, pill count of the medication and monthly urine analysis for the presence of a riboflavin marker. Patients will consume 60 mg riboflavin per day. Riboflavin is rapidly excreted in the urine and is fluorescent when passed under an ultraviolet lamp. In addition, spot checks of blood levels of dilinoleoylphosphatidylcholine (DLPC, the main phosphatidylcholine species of PPC) will validate compliance.

Alcohol intake will be monitored by 3 methods: patient diary, collateral history and monthly blood tests for markers of alcohol consumption (carbohydrate deficient transferrin)(CDT).

Liver biopsies are performed at the end of 3 years and the specimens analyzed by two pathologists who are unaware of the patients' identification and treatment regimen. Fibrosis is the major criterion, with some assessment in additional areas, such as virologic response examined in both drinkers and non-drinkers.

1. Fibrosis: The primary statistical analysis will compare the PPC and placebo groups with regard to changes in fibrosis score from baseline to the value after 36 months of treatment. The primary fibrosis end point is histological with degrees of fibrosis graded on liver biopsy according to Ishak et al (1995). Furthermore, we count the number of α-smooth muscle actin (SMA) expressing stellate cells (Reeves et al, 1996), the principal collagen producing cells. Activation of stellate cells and their transformation to myofibroblast-like cells has been demonstrated in experimental fibrosis (Mak et al, 1984, 1994). Smooth muscle actin α is an actin isoform typical of smooth muscle cells (Skalli et al, 1986), that may be localized in stellate cells of the human liver. Its expression in the stellate cells has been considered an indication of phenotypic modulation of stellate cells to myofibroblasts. In the human liver the appearance of smooth muscle actin α was closely related to the process of hepatic fibrosis (Reeves et al, 1996) and the formation of cirrhotic nodules (Nouchi et al, 1991). In addition, circulating break-down products of collagen or other components of the extracellular matrix (ECM) are being used as markers of liver pathology. These include laminin, the major noncollagenous glycoprotein of basement membranes. Indeed, extracellular basement membranes undergo a continuous turnover and elevation of laminin has been described in the sera of patients with alcoholic liver disease (Niemelä et al. 1988; Sato et al. 1986). Tenascin, a molecule expressed in proliferating ECM, TIMP-1 an inhibitor of the matrix degrading metalloproteinases (MMPs), collagen IV, collagen VI, a molecule that forms filaments between large collagen fibrils, the N-terminal propeptide of procollagen type III (PIIINP), considered a marker of fibrogenesis, hyaluronic acid (HA), an ubiquitous glycosaminoglycan with high extraction by the liver sinusoidal endothelium, and MMP-2. All these have been assessed before as markers of fibrosis, some specifically in patients with chronic hepatitis C (Kasahara et al, 1997; McHutchison et al, 2000; Kojima et la, 2001; Murawaki et al, 2001) but not in subjects who were also drinkers.
2. Sustained virologic response, defined as the absence of plasma HCV RNA a minimum of 24 weeks after antiviral treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (up to 67 years old) are eligible for the study if they are positive for HCV RNA on testing with the polymerase chain reaction (quantitative test), or qualitative test positive if quantitative negative, have undergone a liver biopsy within one year before entry, available for analysis (vide infra) and whose results are consistent with a diagnosis of chronic hepatitis with at least moderate inflammation, a fibrosis score of at least 2/6 according to Ishak et al (1995), and excluding complete cirrhosis. In terms of drinking, the men comprise "abstainers" (less than 12 drinks in the past year), those who drink lightly (1-13 drinks per month) or moderately (4-14 drinks per week) (Dufour, 1999). For women below the age of 50 years, these levels are reduced in half. A drink is defined as: 12 ounces of regular beer, 5 ounces of wine or 1.5 ounces of distilled spirits (80 proof) (Nutrition and Your Health, 1990).

Exclusion Criteria:

-

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2000-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a combined antiviral, antifibrotic and antioxidant treatment on the progression of liver disease in patients with hepatitis C who abstain from alcohol or consume it.

SECONDARY OUTCOMES:
To validate the reliability of various circulating markers as substitute for liver biopsies to indicate the stage of liver pathology and its propensity for progression.

CONTACTS AND LOCATIONS:
Overall Officials: Charles S Lieber, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Bronx VA, The Bronx, New York, United States